CLINICAL TRIAL: NCT06165562
Title: Pressure Supporting Ventilation and Electroencephalography-guided Extubation for Free of Unwanted compLications (PEACEFUL): a Randomised Controlled Trial
Brief Title: Pressure Supporting Ventilation and EEG-guided Emergence for Free of Unwanted Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Associcate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3-2023-0338
Record Dates: First submitted 2023-11-16; First posted 2023-12-11 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Surgery

STUDY DESIGN:
Intervention Model Description: Prospective, single-blinded, parallel-group, randomized clinical study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Patients, medical staff responsible for measuring outcome variables, surgeons, and nurses in the recovery room and wards will be blinded. This blinding approach ensures that both medical staff and patients remain unaware of the assigned group throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure Supporting Ventilation (PSV) and EEG-guided Emergence group (Experimental): Pressure support ventilation will be applied from the start of subcutaneous suture until extubation. At the end of surgery, sevoflurane will be discontinued, and the attending anesthesiologist will perform tracheal extubation after observing the 'zipper opening' pattern on the EEG spectrogram, indicating the patient's recovery of consciousness. For safety reason, extubation will also be guided by the following processed EEG indices thresholds:
  1. 95% spectral edge frequency (SEF) ≥ 23
  2. Patient state index (PSI) ≥ 64
  Interventions: Procedure: PSV; Procedure: EEG-Guidance; Procedure: Spontaneous Respiration
- Conventional Emergence group (Active Comparator): Conventional full-awake extubation will be performed based on the routine practice of our institution. At the end of surgery, sevoflurane will be stopped, and the attending anesthesiologist will lead the emergence process, allowing the patient to breathe spontaneously and providing intermittent manual assistance if necessary. Extubation will be performed when the patient meets the following criteria: obeys commands such as eye-opening or hand-grip, tidal volume > 5 ml/kg, end-tidal carbon dioxide < 45 mmHg, spontaneous respiratory rate 10 to 20 breaths/min.
  Interventions: Procedure: Intermittent Manual Assistance; Procedure: Obey Command; Procedure: Spontaneous Respiration

INTERVENTIONS:
Procedure: PSV — Pressure support ventilation applied from the start of subcutaneous suture until extubation.
  Arms: Pressure Supporting Ventilation (PSV) and EEG-guided Emergence group
Procedure: Intermittent Manual Assistance — Volume-controlled mode during surgery, with intermittent manual assistance from the end of surgery until extubation.
  Arms: Conventional Emergence group
Procedure: EEG-Guidance — Extubation criteria based on EEG findings:Zipper opening pattern observed in the spectrogram 95% spectral edge frequency (SEF) ≥ 23 Patient state index (PSI) ≥ 64
  Arms: Pressure Supporting Ventilation (PSV) and EEG-guided Emergence group
Procedure: Obey Command — Extubation criteria include obeying commands (eye-opening or handgrip).
  Arms: Conventional Emergence group
Procedure: Spontaneous Respiration — Extubation criteria include:
  Tidal volume > 5 ml/kg End-tidal carbon dioxide (ETCO2) < 45 mmHg Spontaneous respiratory rate (RR) 10 to 20 breaths/min

SUMMARY:
This study aims to assess whether pressure supporting ventilation and electroencephalogram (EEG)-guided emergence can reduce airway complications after thyroid surgery compared with conventional emergence. Patients will be randomly assigned to either pressure supporting ventilation and EEG-guided emergence group (intervention group) or conventional emergence group (control group). Co-primary outcomes are the incidence of emergence coughing and lowest percutaneous oxygen saturation (SpO2) after emergence. Secondary outcomes included severity of emergence cough, emergence time, blood pressure and heart rate during emergence, Richmond Agitation-Sedation Scale (RASS) immediately after extubation and upon post-anesthesia care unit (PACU) arrival, incidence of desaturation during PACU stay, hoarseness, sore throat during PACU stay, duration of PACU stay, surgeon satisfaction regarding emergence process, postoperative pain score, and patient satisfaction score regarding emergence process.

DETAILED DESCRIPTION:
Adult patients aged < 40 years scheduled to undergo thyroid surgery will be screened for eligibility. Patients will be randomly allocate to either the intervention group or control group.

* In the intervention group, pressure support ventilation will be applied from the start of subcutaneous suture until extubation. At the end of surgery, sevoflurane will be discontinued, and the attending anesthesiologist will perform tracheal extubation after observing the 'zipper opening' pattern on the EEG spectrogram, indicating the patient's recovery of consciousness. For safety reason, extubation will also be guided by the following processed EEG indices thresholds:

  1. 95% spectral edge frequency (SEF) ≥ 23
  2. Patient state index (PSI) ≥ 64
* In the control group, conventional full-awake extubation will be performed based on the routine practice of our institution. At the end of surgery, sevoflurane will be stopped, and the attending anesthesiologist will lead the emergence process, allowing the patient to breathe spontaneously and providing intermittent manual assistance if necessary. Extubation will be performed when the patient meets the following criteria: obeys commands such as eye-opening or hand-grip, tidal volume > 5 ml/kg, end-tidal carbon dioxide < 45 mmHg, spontaneous respiratory rate 10 to 20 breaths/min.

In both groups, the Oxygen Reserve Index (ORi) will be monitored. Blinded investigator will assess the incidence of emergence coughing and the lowest SpO2 after emergence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged under 40 years who are scheduled to undergo thyroid surgery.

Exclusion Criteria:

* Patients scheduled for radical neck dissection
* Patients scheduled for lymph node biopsy
* Patients with an anticipated difficult airway
* Patients experiencing difficulty during intubation
* Patients with a fasting time not meeting institutional policy
* Patients with a body mass index (BMI) greater than 30 kg/m²
* Patients with sleep apnea
* Pregnant or breastfeeding women
* Patients unable to communicate

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence coughing | During the time period from sevoflurane cessation until 5 minutes after extubation
  Incidence of emergence coughing (defined as coughing during the time period from sevoflurane off until 5 minutes after extubation)
Lowest SpO2 after emergence | During the time period from sevoflurane cessation until post-anesthesia care unit (PACU) discharge, an average of 1 hour
  Lowest SpO2 after emergence (defined as the lowest SpO2 value during the time period from sevoflurane off to post-anesthesia care unit (PACU) discharge)

SECONDARY OUTCOMES:
Severity of Emergence coughing | During the time period from sevoflurane cessation until 5 minutes after extubation.
  The severity of emergence coughing will be assessed using the modified 4-point Minogue scale, with grades assigned as follows: grade 1 (none), grade 2 (mild), grade 3 (moderate), or grade 4 (severe). A higher score indicates a more severe cough.
Incidence and severity of coughing during PACU stay | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  Incidence and severity of coughing during PACU stay evaluated using a modified 4-point Minogue scale.
Emergence time | During the time period from sevoflurane cessation until tracheal extubation, an average of 20 minutes
  Time from sevoflurane cessation until tracheal extubation (minutes)
Time to leave operating room | During the time period from sevoflurane cessation until leaving operating room, an average of 30 minutes
  Time from sevoflurane cessation until leaving operating room
Blood pressure during emergence | during the time period from sevoflurane off until 5 minutes after extubation
  systolic, diastolic, mean blood pressure (mmHg)
Heart rate during emergence | during the time period from sevoflurane off until 5 minutes after extubation
  Heart rate (beats per minute)
Incidence of endotracheal tube biting | During the time period from sevoflurane cessation until tracheal extubation, an average of 20 minutes
  Biting of the endotracheal tube; The investigator will observe whether the patient bites the endotracheal tube or not.
Hypoventilation after extubation (RR <8/min) | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  Hypoventilation defined as Respiratory Rate <8/min
Richmond Agitation-Sedation Scale (RASS) immediately after extubation and upon PACU arrival | RASS will be assessed at two time points; (1) immediately after tracheal extubation, and (2) immediately after PACU arrival
  The Richmond Agitation-Sedation Scale (range : +4 to -5)
Incidence of desaturation during PACU stay | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  Incidence of desaturation
Hoarseness | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  Patients will be specifically asked about the existence of a hoarse voice
Incidence and severity of sore throat | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  Incidence and severity of pain or irritation of the throat.
Duration of PACU stay | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  Duration of PACU stay (minutes)
Surgeon satisfaction regarding emergence process encompassing smoothness/safety/speed | Immediately after the transfer of the patient from operating room to PACU
  Surgeon satisfaction regarding emergence process encompassing smoothness/safety/speed (0: totally unsatisfied, 10: totally satisfied)
Incidence of awareness with recall | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  Patients will be specifically asked whether they experienced intraoperative consciousness, explicit recall of intraoperative events, or the emergence process.
Pain score during PACU stay | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  pain score assessed by numeric rating scale; from 0 (no pain) to 10 (worst pain)
Patient satisfaction score regarding emergence process | During the time period from PACU admission until PACU discharge, an average of 40 minutes
  0: totally unsatisfied, 10: totally satisfied
Incidence of Postoperative hematoma | After operation, through the hospitalization, an average of 3 days.
  hematoma formation
Incidence of wound dehiscence | After operation, through the hospitalization, an average of 3 days.
  dehiscence of the surgical wound
reoperation | After operation, through the hospitalization, an average of 3 days.
  reoperation of thyroid surgery
Oxygen Reserve Index | During the period from sevoflurane cessation until PACU discharge, an average of 1 hour
  Index of the patient's oxygen reserve, with a unit-less scale between 0.00 and 1.00.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Difficult Airway Society Extubation Guidelines Group; Popat M, Mitchell V, Dravid R, Patel A, Swampillai C, Higgs A. Difficult Airway Society Guidelines for the management of tracheal extubation. Anaesthesia. 2012 Mar;67(3):318-40. doi: 10.1111/j.1365-2044.2012.07075.x. PMID 22321104
- [Background] Purdon PL, Pierce ET, Mukamel EA, Prerau MJ, Walsh JL, Wong KF, Salazar-Gomez AF, Harrell PG, Sampson AL, Cimenser A, Ching S, Kopell NJ, Tavares-Stoeckel C, Habeeb K, Merhar R, Brown EN. Electroencephalogram signatures of loss and recovery of consciousness from propofol. Proc Natl Acad Sci U S A. 2013 Mar 19;110(12):E1142-51. doi: 10.1073/pnas.1221180110. Epub 2013 Mar 4. PMID 23487781
- [Background] Jeong H, Tanatporn P, Ahn HJ, Yang M, Kim JA, Yeo H, Kim W. Pressure Support versus Spontaneous Ventilation during Anesthetic Emergence-Effect on Postoperative Atelectasis: A Randomized Controlled Trial. Anesthesiology. 2021 Dec 1;135(6):1004-1014. doi: 10.1097/ALN.0000000000003997. PMID 34610099